CLINICAL TRIAL: NCT00236353
Title: An Open-label Study of the Efficacy and Safety of RISPERDAL Long-acting Microspheres (RISPERDAL CONSTA) Administered Once Monthly in Adults With Schizophrenia or Schizoaffective Disorder
Brief Title: Evaluation of the Efficacy and Safety of Risperidone Injections Given Once a Month to Adults With Schizophrenia or Schizoaffective Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen, LP (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR002830
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-03

CONDITIONS: Schizophrenia; Psychotic Disorders
Keywords: schizophrenia; schizoaffective disorder; long-acting risperidone; intramuscular injection
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
The purpose of this study is to assess the effectiveness and safety of long-acting risperidone given as a once monthly injection to adult patients with schizophrenia or schizoaffective disorder.

DETAILED DESCRIPTION:
Risperidone, taken by mouth on a daily basis, has been an effective treatment for schizophrenia and schizoaffective disorder. Risperidone is also available in a long-acting injectable form so that patients can take their medicine by bi-weekly injections. This study will assess the effectiveness and safety of long-acting risperidone injection given once a month instead of every two weeks (based on previous studies with dosing every 2 weeks). During the four-week lead-in phase, patients will receive one 50-milligram injection every two weeks for two doses. Patients continue to take their prescribed dose of risperidone tablets (from 2 to 6 milligrams per day) for the first 14 days. After the first month, patients will receive one 50-milligram injection once a month for 48 weeks. This dose can be increased to 75 milligrams if patient meets relapse criteria, and is willing to stay in the trial. Patients will be asked questions to help determine how well the monthly injections are working. Laboratory tests (including drug levels), physical examinations and adverse event reporting will be performed to determine the safety of the monthly injections. Risperidone oral tablets, 2 to 6 milligrams per day, for first 2 weeks; long-acting risperidone intramuscular injections, 50 mg in 2 milliliters of liquid, every 2 weeks for 1 month, then injections once a month for 48 weeks. Monthly injection dose may be increased to 75 mg in 2-mL if needed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder
* stable with respect to disease symptoms and other medical conditions
* stable on antipsychotic therapy with oral risperidone 2 to 6 milligrams per day for 8 weeks before study
* if female, using birth control.

Exclusion Criteria:

* Hospitalized within 8 weeks of beginning the study
* at risk to self or others
* presence of liver or kidney damage
* use of oral antipsychotic drugs other than risperidone within the past 8 weeks, of injected antipsychotics within the past 6 months, of long-acting risperidone in an earlier study, of investigational drugs within the past 30 days, or of electroconvulsive therapy within the past 12 months
* pregnant or breast-feeding
* if female, not using birth control
* abusing drugs or alcohol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2002-05; Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Effectiveness measured by incidence of symptom reoccurrence (relapse) in 1 year.

SECONDARY OUTCOMES:
Effectiveness assessed by the Clinical Global Impression Scale, Positive and Negative Syndrome Scale; safety scales are for: Extrapyramidal Symptom Rating, Abnormal Involuntary Movement, and Dickson-Glazer Sexual Functioning Inventory, and adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Janssen, LP Clinical Trial, Study Director — Janssen, LP

REFERENCES:
- [Derived] Uchida H, Mamo DC, Kapur S, Labelle A, Shammi C, Mannaert EJ, Mann SW, Remington G. Monthly administration of long-acting injectable risperidone and striatal dopamine D2 receptor occupancy for the management of schizophrenia. J Clin Psychiatry. 2008 Aug;69(8):1281-6. doi: 10.4088/jcp.v69n0811. PMID 18642974
- See also: An Open-Label Study of the Efficacy and Safety of RISPERDAL� Long-Acting Microspheres (RISPERDAL� CONSTA�) administered once monthly in Adults with Schizophrenia or Schizoaffective Disorder — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=346&filename=CR002830_CSR.pdf